CLINICAL TRIAL: NCT06275477
Title: 68Gallium-FAPI PET/CT Imaging in Chronic Inflammatory and Fibrotic Diseases
Acronym: PARADISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC23.0029
Record Dates: First submitted 2024-01-29; First posted 2024-02-23 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Disease

STUDY DESIGN:
Intervention Model Description: This is a single-center, descriptive and analytical pilot study, which will be implemented in 13 distinct and independent populations of patients with chronic inflammatory and/or fibrosing disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ga68-FAPI46 TEP scan (Experimental): In addition to the usual routine care, the study adds the performance of a [68Ga] Ga-FAPI PET/CT scan
  Interventions: Diagnostic Test: 68Ga-FAPI46

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI46 — Depending on the situation, it is planned that this evaluation will be transversal (performing [68Ga] Ga-FAPI PET/CT at baseline) or longitudinal (performing [68Ga] Ga-FAPI PET/CT at baseline and at 3/6 months for patients benefiting from an intensification of therapeutic management at inclusion).

SUMMARY:
This single-center pilot study is designed to explore the preliminary utility of the [68Ga] Ga-FAPI imaging agent in positron emission tomography (PET) combined with computed tomography (CT) for a range of chronic inflammatory and fibrosing diseases. The study focuses on the potential of [68Ga] Ga-FAPI, a novel radiotracer targeting Fibroblast Activation Protein (FAP), to improve diagnostic accuracy in various medical conditions. Thirteen distinct clinical situations have been selected for this investigation, including rheumatoid arthritis, liver fibrosis, and systemic lupus, among others. This approach aims to ascertain the value of further clinical development in each area and refine the use of this imaging modality in routine care for both initial evaluation and ongoing monitoring of these diseases.

DETAILED DESCRIPTION:
[68Ga] Ga-FAPI is an innovative radiotracer in positron emission tomography (PET) coupled to scanner (CT: computed tomography). It targets the membrane glycoprotein FAP (Fibroblast Activation Protein), a specific surface marker of activated fibroblasts, these constituting one of the main populations of the tumor microenvironment. This radiotracer is the subject of a major development program in the field of oncology and hematologic malignancies. In many cancers, preliminary data suggest, in terms of diagnostic performance, the superiority of [68Ga] Ga-FAPI over the reference evaluation modality carried out with [18F] F-FDG. These results make it possible to consider, in the medium term, the integration of this imaging modality into routine care, for the initial evaluation and monitoring of certain tumor pathologies.

If oncology and hematology constitute the most obvious areas of application of [68Ga] Ga-FAPI, other areas of potential use were quickly mentioned, due to the involvement of activated fibroblasts in the processes. remodeling of the extracellular matrix and tissue repair in general, beyond tumor pathologies. Non-exhaustively, the potential interest of the radiotracer is thus suggested in the characterization of benign tumor pathologies, in the evaluation of ischemic tissues, in chronic inflammatory diseases and in fibrosing diseases. Numerous preliminary data show that it is relevant to develop knowledge concerning the contribution of [68Ga] Ga-FAPI to the evaluation of numerous benign pathologies.

It is in this general context that this single-center pilot study project falls, the general objective of which is to determine the preliminary interest of this imaging modality in different chronic inflammatory and/or fibrosing diseases. The pathologies included in this project were selected by taking into account the concomitant presence of unmet medical needs in terms of disease assessment and recognized local clinical research expertise in the area concerned. On these bases, 13 distinct clinical situations were selected, intended to enable the production of pilot data. This approach will be able to determine the interest in continuing clinical development in each area and will help to specify the modalities.

The 13 clinical situations selected for this pilot study are:

* Rheumatoid arthritis
* Spondyloarthritis
* Inflammatory enterocolopathies
* Liver fibrosis
* Fibrosing interstitial lung disease
* Systemic sarcoidosis
* Polymyalgia rheumatica and giant cell arteritis
* Primary Sjögren's syndrome
* Systemic scleroderma
* Systemic lupus
* Inflammatory myopathies
* Primary or secondary myelofibrosis
* Other orphan systemic diseases

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over.
* Affected by one of the pathologies concerned by the study (see Table 4)
* Satisfying the consensus classification criteria for the pathology (Table 3).
* Satisfying the corresponding clinical situation (Table 3).
* Negative urine pregnancy test for women of childbearing age.
* Affiliated with or benefiting from social security.
* Informed consent (personally dated and) signed by the participant or any representatives (impartial witness/trusted person).

Exclusion Criteria:

* Patients unable to consent.
* Incapacitated adults.
* Pregnant or breastfeeding women.
* Patients refusing to participate in research.
* Known active cancer.
* Women of childbearing potential unwilling to use appropriate contraception (definitions given in Annex 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-09-21 (Estimated); Study Completion 2027-09-21 (Estimated)

PRIMARY OUTCOMES:
PET uptake intensity | Month 0
  Describe the sites and intensity of fixation of [68Ga] Ga-FAPI PET/CT measured by the Standardized uptake value (SUV) max on the examination performed at M0 in the 13 targeted chronic inflammatory and/or fibrosing diseases.

SECONDARY OUTCOMES:
[68Ga]Ga-FAPI PET/CT - Pathology evaluation correlation | Month 0
  - Measurement of PET fixation intensity
[68Ga]Ga-FAPI PET/CT - Pathology evaluation correlation | Month 0
  - Measurement of the pathology-specific reference score (if applicable)
[68Ga]Ga-FAPI PET/CT - Pathology evaluation correlation | Month 3
  - Measurement of PET fixation intensity
[68Ga]Ga-FAPI PET/CT - Pathology evaluation correlation | Month 3
  - Measurement of the pathology-specific reference score (if applicable)
[68Ga]Ga-FAPI PET/CT - Pathology evaluation correlation | Month 6
  - Measurement of PET fixation intensity
[68Ga]Ga-FAPI PET/CT - Pathology evaluation correlation | Month 6
  - Measurement of the pathology-specific reference score (if applicable)
[68Ga]Ga-FAPI PET/CT - Others pathology evaluation correlation | Month 0
  - Measurement of PET uptake intensity
[68Ga]Ga-FAPI PET/CT - Others pathology evaluation correlation | Month 0
  - Measurement of other pathology-specific assessment scores (if applicable)
[68Ga]Ga-FAPI PET/CT - Others pathology evaluation correlation | Month 3
  - Measurement of PET uptake intensity
[68Ga]Ga-FAPI PET/CT - Others pathology evaluation correlation | Month 3
  - Measurement of other pathology-specific assessment scores (if applicable)
[68Ga]Ga-FAPI PET/CT - Others pathology evaluation correlation | Month 6
  - Measurement of PET uptake intensity
[68Ga]Ga-FAPI PET/CT - Others pathology evaluation correlation | Month 6
  - Measurement of other pathology-specific assessment scores (if applicable)
[68Ga]Ga-FAPI PET/CT - Biomarkers correlation | Month 0
  - Measurement of PET fixation intensity
[68Ga]Ga-FAPI PET/CT - Biomarkers correlation | Month 0
  - Measurement of pathology-specific biological markers (if applicable). Biomarkers are specific to the pathologies studied (may include: CRP, Hb, Albumin, CRP, fecal calprotectin, IgG, native anti-DNA, proteinuria, CPK, ECA...).
[68Ga]Ga-FAPI PET/CT - Biomarkers correlation | Month 3
  - Measurement of PET fixation intensity
[68Ga]Ga-FAPI PET/CT - Biomarkers correlation | Month 3
  - Measurement of pathology-specific biological markers (if applicable). - Measurement of pathology-specific biological markers (if applicable). Biomarkers are specific to the pathologies studied (may include: CRP, Hb, Albumin, CRP, fecal calprotectin, IgG, native anti-DNA, proteinuria, CPK, ECA...).
[68Ga]Ga-FAPI PET/CT - Biomarkers correlation | Month 6
  - Measurement of PET fixation intensity
[68Ga]Ga-FAPI PET/CT - Biomarkers correlation | Month 6
  - Measurement of pathology-specific biological markers. - Measurement of pathology-specific biological markers (if applicable). Biomarkers are specific to the pathologies studied (may include: CRP, Hb, Albumin, CRP, fecal calprotectin, IgG, native anti-DNA, proteinuria, CPK, ECA...).
[68Ga]Ga-FAPI PET/CT - Functional parameters correlation | Month 0
  - Measurement of PET fixation intensity
[68Ga]Ga-FAPI PET/CT - Functional parameters correlation | Month 0
  - Measurement of pathology-specific functional parameters.
[68Ga]Ga-FAPI PET/CT - Functional parameters correlation | Month 3
  - Measurement of PET fixation intensity
[68Ga]Ga-FAPI PET/CT - Functional parameters correlation | Month 3
  - Measurement of pathology-specific functional parameters
[68Ga]Ga-FAPI PET/CT - Functional parameters correlation | Month 6
  - Measurement of PET fixation intensity
[68Ga]Ga-FAPI PET/CT - Functional parameters correlation | Month 6
  - Measurement of pathology-specific functional parameters.
[68Ga]Ga-FAPI PET/CT - Imaging characteristics correlation | Month 0
  - Measurement of PET uptake intensity
[68Ga]Ga-FAPI PET/CT - Imaging characteristics correlation | Month 0
  - Measurement of pathology-specific imaging characteristics.
[68Ga]Ga-FAPI PET/CT - Imaging characteristics correlation | Month 3
  - Measurement of PET uptake intensity
[68Ga]Ga-FAPI PET/CT - Imaging characteristics correlation | Month 3
  - Measurement of pathology-specific imaging characteristics.
[68Ga]Ga-FAPI PET/CT - Imaging characteristics correlation | Month 6
  - Measurement of PET uptake intensity
[68Ga]Ga-FAPI PET/CT - Imaging characteristics correlation | Month 6
  - Measurement of pathology-specific imaging characteristics.
[68Ga] Ga-FAPI PET/CT parameters evolution | Month 0
  Describe the evolution of [68Ga] Ga-FAPI PET/CT parameters between M0 and M3 (Ki mean, Ki max (ml/min/100ml))
[68Ga] Ga-FAPI PET/CT parameters evolution | Month 3
  Describe the evolution of [68Ga] Ga-FAPI PET/CT parameters between M0 and M3 (Ki mean, Ki max (ml/min/100ml))
[68Ga] Ga-FAPI PET/CT / [18F] F-FDG PET/CT comparison | Month 0
  - Measurement of the fixation intensity in PET/CT with [68Ga] Ga-FAPI and measurement of the fixation intensity in PET/CT with [18F] F-FDG at M0
[68Ga] Ga-FAPI PET/CT kinetic | Month 0
  • Evaluation of the kinetics of uptake of the tracer [68Ga] Ga-FAPI in PET according to the different pathologies and their phenotypic characteristics (Distribution Volume (DV) mean, DV max (%))
[68Ga] Ga-FAPI PET/CT kinetic | Month 3
  • Evaluation of the kinetics of uptake of the tracer [68Ga] Ga-FAPI in PET according to the different pathologies and their phenotypic characteristics (Distribution Volume (DV) mean, DV max (%))
[68Ga] Ga-FAPI PET/CT kinetic | Month 6
  • Evaluation of the kinetics of uptake of the tracer [68Ga] Ga-FAPI in PET according to the different pathologies and their phenotypic characteristics (Distribution Volume (DV) mean, DV max (%))

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Undecided